CLINICAL TRIAL: NCT04104581
Title: Measuring Daily Grain Intake Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HS64 Daily Grain
Record Dates: First submitted 2019-08-28; First posted 2019-09-26 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Placebo Comparator): Volunteers will consume a diet in which all grain foods are made from refined grains.
  Interventions: Other: Control Refined Grain Diet
- Low Whole Grain Oat Diet (Experimental): Volunteers will consume a diet with a low level of whole grain oat incorporated into some of the foods.
  Interventions: Other: Low Whole Grain Oat Diet
- High Whole Grain Oat Diet (Experimental): Volunteers will consume a diet with a high level of whole grain oat incorporated into some of the foods.
  Interventions: Other: High Whole Grain Oat Diet
- Low Whole Grain Wheat Diet (Experimental): Volunteers will consume a diet with a low level of whole grain wheat incorporated into some of the foods.
  Interventions: Other: Low Whole Grain Wheat Diet
- High Whole Grain Wheat Diet (Experimental): Volunteers will consume a diet with a high level of whole grain wheat incorporated into some of the foods.
  Interventions: Other: High Whole Grain Wheat Diet

INTERVENTIONS:
Other: Control Refined Grain Diet — Subjects will be fed the average American diet except it will be free of whole grains
  Arms: Control
Other: Low Whole Grain Oat Diet — Subjects will be fed the average American diet with addition of a low level of whole grain oats
  Arms: Low Whole Grain Oat Diet
Other: High Whole Grain Oat Diet — Subjects will be fed the average American diet with addition of a high level of whole grain oats
  Arms: High Whole Grain Oat Diet
Other: Low Whole Grain Wheat Diet — Subjects will be fed the average American diet with addition of a low level of whole grain wheat
  Arms: Low Whole Grain Wheat Diet
Other: High Whole Grain Wheat Diet — Subjects will be fed the average American diet with addition of a high level of whole grain wheat
  Arms: High Whole Grain Wheat Diet

SUMMARY:
The primary objective of this study is to identify markers of daily whole grain oat and whole grain wheat intake in humans.

DETAILED DESCRIPTION:
The aim of this study is to identify compounds that are found in blood and urine and are derived from repeated daily consumption of whole grain oat or whole grain wheat intake so that epidemiological studies can be conducted to provide more accurate associations between whole grain intake and health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 - 75 years
* non smokers

Exclusion Criteria:

* Body weight less than 110 lbs.
* Have a body mass index below 19 or above 38 kg/m2
* Known (self-reported) allergy or adverse reaction to study foods
* Women who have given birth during the previous 12 months or who are pregnant/lactating or who plan to become pregnant during the study
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease), Crohn's disease, diabetes, or metabolic disorders that may interfere with the study
* History of certain cancer diagnosis or treatment in the last 3 years
* Smoking or use of tobacco products in the past 6 months
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Use of certain medications or supplements (prescription or over-the-counter) that may interfere with the study objectives, including blood thinning medications
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Identification of unknown blood biomarkers of grain intake | Day 1 of Period 1 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 1 of Period 2 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 1 of Period 3 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 1 of Period 4 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 1 of Period 5 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 8 of Period 1 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 8 of Period 2 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 8 of Period 3 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 8 of Period 4 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 8 of Period 5 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 15 of Period 1 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 15 of Period 2 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 15 of Period 3 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 15 of Period 4 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Identification of unknown blood biomarkers of grain intake | Day 15 of Period 5 (period = 15 days)
  Metabolomic analysis of blood samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined

SECONDARY OUTCOMES:
Identification of unknown urinary biomarkers of grain intake | Day 1, 8, and 15 of each of the 5 fifteen day diet periods
  Metabolomic analysis of urine samples will be conducted; the selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight will be determined
Characterization of fecal microbiota | Day 1, 8, and 15 of each of the 5 fifteen day diet periods
  Fecal samples will be analyzed for microbiota
Blood Glucose | Day 1 and 15 of each of the 5 fifteen day diet periods
  Fasting blood glucose will be measured in mg/dL
Blood Insulin | Day 1 and 15 of each of the 5 fifteen day diet periods
  Fasting blood insulin will be measured in uIU/mL
Blood Triglycerides | Day 1 and 15 of each of the 5 fifteen day diet periods
  Fasting blood triglycerides will be measured in mg/dL
Blood Non-Esterified Fatty Acids | Day 1 and 15 of each of the 5 fifteen day diet periods
  Fasting blood non esterified fatty acids will be measured in mEQ/L

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Li Y, Novotny JA, Baer D, Hu Y, Sun Q, Zhang S, Sang S. Betainized metabolites as biomarkers of whole grain wheat, not oat: insights from controlled crossover pharmacokinetic and daily feeding studies. Am J Clin Nutr. 2025 Dec 19:101139. doi: 10.1016/j.ajcnut.2025.101139. Online ahead of print. PMID 41423132